CLINICAL TRIAL: NCT05056116
Title: A Safety and Efficacy Study of Surufatinib Combination With Toripalimab in Patients With Recurrent Biliary Tract Cancer : a Phase Ⅱ Study
Brief Title: A Safety and Efficacy Study of Surufatinib Combination With Toripalimab in Patients With Recurrent Biliary Tract Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Affiliated Hospital of Xuzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMPL-012-SPRING-B101
Record Dates: First submitted 2021-09-15; First posted 2021-09-24 (Actual); Last update posted 2021-12-27 (Actual); Status verified 2021-12

CONDITIONS: Biliary Tract Cancer
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — surufatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Biliary Tract Cancer (Experimental): Surufatinib 250mg/Toripalimab 240mg
  Interventions: Drug: Surufatinib Toripalimab

INTERVENTIONS:
Drug: Surufatinib Toripalimab — Surufatinib at a dose of 250mg Qd, with humanized anti-PD-1 monoclonal antibody Toripalimab injected intravenously 240mg per 3 weeks until disease progresses or unacceptable tolerability occurs.
  Other Names: Surufatinib/JS001

SUMMARY:
A Phase Ⅱ, open-label, single-arm study to assess the safety, tolerability, and efficacy of Surufatinib Combination With Toripalimab in Patients With Recurrent Biliary Tract Cancer.

DETAILED DESCRIPTION:
A Phase 2, open-label, single-arm study to assess the safety, tolerability, and efficacy of Surufatinib Combination With Toripalimab in Patients With Recurrent Biliary Tract Cancer (intrahepatic or extrahepatic cholangiocarcinoma, gallbladder cancer).

ELIGIBILITY:
Inclusion Criteria:

1. Male and Female aged between 18 and 75 years are eligible; Provision of written Informed Consent Form (ICF) prior to any study specific procedures;
2. Advanced (unresectable) or metastatic biliary carcinomas that have been histologically or cytologically confirmed include intrahepatic or extrahepatic carcinoma of the bile duct, carcinoma of the gallbladder, and carcinoma of the ampullary of fatt, and have been histologically confirmed as adenocarcinoma;
3. Patients who have previously received disease progression or toxic side effects after first-line systemic chemotherapy are not tolerated;The standard first-line chemotherapy regimen was defined as a two-drug combination regimen of gemcitabine plus cisplatin, gemcitabine plus gio, or capecitabine plus oxaliplatin.Failure of first-line standard chemotherapy was defined as progression of disease during treatment or within 6 months after the last treatment;Or the toxic side effects of the treatment process are intolerable;
4. Presence of at least one measurable target lesion for further evaluation according to RECIST criteria;
5. Patients who had previously received A VEGF or VEGFR-targeted drug required progression 4 months after the last dose;
6. No systemic antitumor therapy in 4 weeks;
7. The patient has no evidence of biliary obstruction unless the obstruction is controlled by local treatment or the patient is decompressed by endoscopic or percutaneous stenting, and bilirubin is subsequently reduced to below the upper limit of 1.5x normal (ULN);
8. Eastern Cooperative Oncology Group (ECOG) performance status 0-1;Predicted survival ≥3 months;
9. Screening laboratory values must meet the following criteria (within past 14 days):

   * neutrophils ≥1.5×109/L ;
   * platelets ≥9g/dL；
   * hemoglobin ≥ 9.0 g/dL;
   * albumin≥3g/dL；
   * total bilirubin ≤ 1.5 x upper limit of normal (ULN); aspartic transaminase (AST) and alanine transaminase (ALT) ≤ 2.5 x ULN without, and ≤ 5 x ULN with hepatic metastasis; serum creatinine ≤1.5╳ULN;
10. Voluntary enrollment, good compliance, can cooperate with the experiment observation, and signed a written informed consent;
11. Males or female of childbearing potential must: agree to use using a reliable form of contraception (eg, oral contraceptives, intrauterine device, control sex desire, double barrier method of condom and spermicidal) during the treatment period and for at least 6 months after the last dose of study drug.

Exclusion Criteria:

1. Prior treatment with Surufatinib,or other antiangiogenic drugs were used within 6 months;
2. Prior antitumor therapy with chemotherapy, radical radiation therapy ，biological immunotherapy，targeted therapy within 4 weeks.
3. Prior participation in other clinical trials not approved or listed in China within past 4 weeks；
4. Prior major surgery within past 4 weeks (diagnostic surgery excluded);
5. International standardized ratio (INR) >1.5 or partially activated prothrombin time (APTT) >1.5×ULN;
6. Clinically significant severe electrolyte abnormality judged by investigator ;
7. Hypertension that is not controlled by the drug, and is defined as: SBP≥140 mmHg and/or DBP≥90 mmHg;
8. Currently suffering from poorly controlled diabetes (after regular treatment, fasting plasma glucose concentration ≥10mmol/L);
9. The patient currently has disease or condition that affects the absorption of the drug, or the patient cannot be administered orally;
10. Digestive tract disease such as gastric and duodenal active ulcer, ulcerative colitis or unresected tumor, or other conditions determined by the investigator that may cause gastrointestinal bleeding and perforation;
11. Evidence of bleeding tendency or history within 3 months, or thromboembolic event (including a stroke event and/or a transient ischemic attack) occurred within 12 month;
12. Cardiovascular disease of significant clinical significance (myocardial infarction, unstable arrhythmia or unstable angina ，Coronary Artery Bypass Grafting within past 6 months,)；
13. Had other malignant tumors in the past 5 years (except for basal cell carcinoma or squamous cell carcinoma, cervical carcinoma in situ that have been effectively controlled);
14. Active or uncontrolled severe infection (≥CTCAE2 infection);
15. Positive tests for HIV, HCV, HBsAg or HBcAb with positive test for HBV DNA (>2000IU/ml);
16. Evidence with active CNS disease or previous brain metastases;
17. The toxicity associated with previous anti-tumor treatment has not recovered to ≤CTCAE1, except for peripheral neurotoxicity and alopecia ≤CTCAE2 caused by oxaliplatin;
18. Pregnant or nursing;
19. Transfusion therapy, blood products and hematopoietic factors, such as albumin and granulocyte colony stimulating factor (G-CSF), had been received within 14 days before enrollment;
20. Tumor involving skin and/or pharyngeal mucosa with ulceration;
21. Patients with a history of psychotropic drug abuse and unable to quit or with mental disorders;
22. Any other disease, with clinical significance of metabolic abnormalities, abnormal physical examination or laboratory abnormalities, according to researchers, there is reason to doubt is not suitable for the use of study drugs in patients with a disease or condition (such as have a seizure and require treatment), or will affect the interpretation of results, or make the patients at high risk.
23. Routine urine indicated that urine protein ≥2+, and the 24-hour urine protein volume >1.0g;
24. Underlying medical condition that, in the Investigator's opinion, would increase the risks of study drug administration or obscure the interpretation of toxicity determination or adverse events.
25. Prior receipt of any anti-PD-1 /PD-L1/PD-L2 antibody or anti-cytotoxic T lymphocyte associated antigen-4 (CTLA-4) antibody or any other antibody acting on T cell co-stimulation or checkpoint pathway (e.g. OX40, CD137, etc.)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Objective response rate(ORR) | up to 24 months
  The number of cases in which tumor size is reduced to PR or CR / the total number of evaluable cases (%). In the event of PR or CR, the subjects should confirm it no less than 4 weeks after the first evaluation. CT/MRI will be performed every 2 cycles of treatment by RECIST 1.1(each cycle is 21 days))

SECONDARY OUTCOMES:
Progression-free survival (PFS) | up to 12 months
  To assess the efficacy of Surufatinib Combination With Toripalimab in Patients With Recurrent Biliary Tract Cancer, patients by assessment of progression free survival (PFS) using Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1).
Overall survival (OS) | up to 36 months
  The time interval between the start date of study drug and the date of death (any cause).

CONTACTS AND LOCATIONS:
Overall Officials: Renhao Wang, MD, Principal Investigator — The Affiliated Hospital of Xuzhou Medical University; Bin Zhang, MD, Principal Investigator — The Affiliated Hospital of Xuzhou Medical University
Locations (1):
- The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu, China